CLINICAL TRIAL: NCT01552512
Title: Randomized Control Trial of Complementary Food to Prevent Undernutrition Among At-Risk Infants in Fort San Michel, Haiti
Brief Title: Nutributter Programming to Prevent Undernutrition: an Evaluation
Acronym: NPPU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: University of California, Davis (Other); World Bank (Other); United Nations World Food Programme (WFP) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FSM-001-201101760
Record Dates: First submitted 2012-02-15; First posted 2012-03-13 (Estimated); Last update posted 2018-08-06 (Actual); Status verified 2018-08

CONDITIONS: Undernutrition
Keywords: Stunting; Hidden Hunger; Diarrhea; Vitamin A Deficiency
MeSH Terms: conditions — Malnutrition; Growth Disorders; Diarrhea; Vitamin A Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- MSPP Integrated Package (No Intervention): Participants in this arm only receive the standard care offered by the Ministry of Health (MSPP)called the Integrated Package. During the trial, they do not receive Nutributter.
- Nutributter 3 Months, Integrated Package (Experimental): Participants receive a one-month supply for the first 3 months of the 6-month trial in addition to the Integrated Package.
  Interventions: Dietary Supplement: Nutributter Program; Other: Integrated Package
- Nutributter 6 Months, Integrated Package (Experimental): Participants receive a one-month supply for each month of the 6-month trial in addition to the Integrated Package.
  Interventions: Dietary Supplement: Nutributter Program; Other: Integrated Package

INTERVENTIONS:
Dietary Supplement: Nutributter Program — Nutributter is a ready-to-use nutritional supplement that provides all vitamins and minerals required for healthy growth of infants 6 to 12 months of age. The paste is packaged in 20 gram sachets. One sachet corresponds to the recommended daily dose for a child.
  Other Names: Nutriset
  Arms: Nutributter 3 Months, Integrated Package; Nutributter 6 Months, Integrated Package
Other: Integrated Package — The integrated package of services are provided through the Haitian Ministry of Health and includes childhood vaccinations, family planning messages, diarrhea prevention and control (e.g. water purification methods, promotion of positive sanitation and hygiene practices such as hand washing), and the promotion of positive child feeding practices (e.g. exclusive breastfeeding for six months; increased frequency of complementary feeding; and dietary diversity).
  Arms: Nutributter 3 Months, Integrated Package; Nutributter 6 Months, Integrated Package

SUMMARY:
This randomized, controlled effectiveness study examines Nutributter programming within an integrated package of maternal and child health services offered by Haiti's Ministry of Health (MSPP) to prevent undernutrition among young children in Haiti. The aim of the process evaluation is to better understand the uptake of Nutributter® as a complementary food in the diets of young children and its feasibility and acceptability as part of MSPP's package of services. This project is being carried out at a public hospital in Fort San Michel, an impoverished community outside of Cap Haitien, Haiti.

ELIGIBILITY:
Inclusion Criteria:

* Infants 6 to 12 months old
* Lives in Fort San Michel

Exclusion Criteria:

* Moderately or severely malnourished
* Peanut allergy

Ages: 6 Months to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1228 (Actual)
Dates: Start 2011-06 (Actual); Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Change in Length for Age | Once per month for 6 months, then once after 12 months.
  Length (measured in centimeters) for age is an indicator of stunting, an outcome of chronic undernutrition during the first 2 years of life. Because our primary purpose is to prevent undernutrition, we are highly interested in this measurement.

SECONDARY OUTCOMES:
Change in Weight for Height | Once per month for 6 months, then once after 12 months
  Weight (measured in kilograms) for height (measured in centimeters) is an indicator of moderate to severe acute malnutrition and if an infant is underweight, she/he could require immediate medical attention. We therefore weigh each participant to assess their current health status in this regard.

CONTACTS AND LOCATIONS:
Overall Officials: Lora Iannotti, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Hopital Fort San Michel, Cap-Haïtien, Haiti

REFERENCES:
- [Derived] Iannotti LL, Dulience SJ, Green J, Joseph S, Francois J, Antenor ML, Lesorogol C, Mounce J, Nickerson NM. Linear growth increased in young children in an urban slum of Haiti: a randomized controlled trial of a lipid-based nutrient supplement. Am J Clin Nutr. 2014 Jan;99(1):198-208. doi: 10.3945/ajcn.113.063883. Epub 2013 Nov 13. PMID 24225356